CLINICAL TRIAL: NCT02025920
Title: Title in Norwegian: Sunn og Frisk. En Studie av Helseeffekter av Fiskeinntak i Overvektige Voksne (FINS)
Brief Title: Project Healthy Eating in Adults. A Study on the Health Effects of Fish Intake in Overweight Adults (FINS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: The Fisheries and Aquaculture Industry Research Fund (Other)
Responsible Party: Principal Investigator, Oddrun Anita Gudbrandsen, Researcher, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013/558
Record Dates: First submitted 2013-12-17; First posted 2014-01-01 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Overweight or Obese Adults; Healthy
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Salmon Group (Experimental): Participants will eat 150g salmon for dinner, 3 times per week for 12 weeks
  Interventions: Other: Salmon Group
- Cod Group (Experimental): Participants will eat 150g cod for dinner, 3 times per week for 12 weeks
  Interventions: Other: Cod Group
- Meat Group (Active Comparator): Participants will eat 150g mixed meat for dinner, 3 times per week for 12 weeks
  Interventions: Other: Meat Group

INTERVENTIONS:
Other: Salmon Group
  Arms: Salmon Group
Other: Cod Group
  Arms: Cod Group
Other: Meat Group
  Arms: Meat Group

SUMMARY:
It has previously been observed that increased fish intake improves the metabolic health of overweight and obese adults, and animal protein improved metabolic health of obese rats. In this project the investigators will investigate whether increased intake of fish or meat improves metabolic health in overweight/obese adults aged 20-55 years when replacing processed food. The hypothesis is that increased intake of unprocessed fish or meat will improve metabolic health in adults as measured by glucose tolerance, lipid metabolism and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 27
* 20-55 years
* healthy

Exclusion Criteria:

* diagnosed diseases such as diabetes, CVD, intestinal diseases, arthritis
* prescription medications affecting the metabolism of glucose, lipids or the immune system
* use of supplements containing long chain n-3 fatty acids
* high intake of fish
* food allergy

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Changes in metabolic status (glucose, lipids, inflammation) | Baseline and end of intervention (12 weeks)
  The effects of fish intake on glucose homeostasis, lipid metabolism and inflammation will be assessed.

SECONDARY OUTCOMES:
Changes in plasma concentrations of amino acids and their metabolites | Baseline and end of intervention (12 weeks)
Changes in plasma concentrations of vitamins | Baseline and end of intervention (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Oddrun A Gudbrandsen, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Norway